CLINICAL TRIAL: NCT06093724
Title: Prospective Imaging Assessment of Perineo-pelvic Static's Evolution After Sexual Reassignment Surgery in MtF Transgender Patient, by Peno-scrotal Inversion Vaginoplasty Technique (TRANSPELV)
Acronym: TRANSPELV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 87RI23_005-TRANSPELV
Record Dates: First submitted 2023-09-08; First posted 2023-10-23 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Transgenderism
Keywords: MtF, transgender, vaginoplasty, penoscrotal inversion, MRI
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anatomy reorganization after vaginoplasty in transgender women (MtF) (Experimental): The research consists of adding to the usual MtF transgender patient undergoing vaginoplasty care course, static and dynamic perineo-pelvic MRI before, and at 6 and 24 months. The aim is to assess perineo-pelvic static's evolution, based on the appearance of a rectocele.
  Interventions: Diagnostic Test: Static and dynamic perineo-pelvic MRI

INTERVENTIONS:
Diagnostic Test: Static and dynamic perineo-pelvic MRI — Static and dynamic perineo-pelvic MRI before surgery, and at 6 and 24 months after surgery.

SUMMARY:
The research consists of adding to the usual MtF transgender patient undergoing vaginoplasty care course, static and dynamic perineo-pelvic MRI before, and at 6 and 24 months. The aim is to assess perineo-pelvic static's evolution, based on the appearance of a rectocele.

DETAILED DESCRIPTION:
Transgender people are estimated to be about 0,3 to 1 % of general population, and MtF reassignment surgery is raising. Vaginoplasty is not always necessary, but is usually an important step into gender transition. In France, surgical techniques' gold-standard is the peno-scrotal inversion vaginoplasty, which consists in the creation of a neo-vagina with peno-scrotal skin graft. Genital, perineum and pelvic anatomy is modified, without knowing in advance about functional and aesthetic results. MRI is the best way to assess soft tissue anatomy in the pelvis. Though, only few studies have assessed pre and post-operative imaging in patients undergoing vaginoplasty, and none have been prospective, neither have assessed the risk of rectocele. The issue is legitimate, because the surgery weakens elements of pelvic fixity, and fixity issues can appear secondarily.

MtF transgender patients operated for a vaginoplasty are undergoing static and dynamic MRI before the surgery, at 6 and at 24 post-operative months. We look after the appearance of a rectocele and it's evolution in time, as criteria for the assessment of pelvic fixity.

Follow-up is composed of several consultations including post-operative MRI, but also clinical measures, census of post-operative issues, and questionnaires for the assessment of secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient admitted in urology ward at Limoges' University Hospital for MtF sexual reassignment surgery by vaginoplasty
* Patient affiliated or benefitting from a social security system
* Patient free, informed, written and signed consent

Exclusion Criteria:

* Patient admitted for vulvoplasty surgery
* Patient admitted for second vaginoplasty surgical gesture
* Contraindication of realizing an MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient admitted in urology ward at Limoges' University Hospital for MtF sexual reassignment surgery by vaginoplasty
Enrollment: 50 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-09-08 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Measurement comparison of the rectal bulge's size and classification | 6 months and 24 months
  Comparison and classification by pre-operative and post-operative MRI

SECONDARY OUTCOMES:
Rectocele | 6 months and 24 months
  Describe the rectocele's mean size and it's progress
Rectocele | 6 months and 24 months
  Describe the rectocele size's progress by class
Reproducibility in the rectocele's measurement | 6 months and 24 months
  Evaluate intra and inter-operator reproducibility in the rectocele's measurement
Symptomatology pelvic fixity | 6 months and 24 months
  Evaluate correlation between symptomatology and the rectocele assessment
Factors pelvic fixity | 6 months and 24 months
  Evaluate correlation between factors and the rectocele assessment
Skin-graft's neo-vagina's sizes | 6 months and 24 months
  Evaluate correlation between the skin-graft's size in cm² and the neo-vagina's sizes (lenght, width) in cm
Imaging measures | 6 months and 24 months
  Evaluate modifications of imaging measures size in cm² and the neo-vagina's sizes (lenght, width) in cm
Urinary quality | 6 months and 24 months
  Evaluate evolution of unrinary quality of life with Urinary Symptom Profile (USP) score, from 0 (best) to 39 (worst)
Self-imaging | 6 months and 24 months
  Evaluate evolution of self-imaging with Body Image (BI-1) score, from 30 (no change) to 150 (change) ; and Female Genital Self-Image Scale (FGSIS) score, from 7 (worst) to 28 (best)
Sexual quality | 6 months and 24 months
  Evaluate evolution of sexual quality of life with Operated Male-to-Female Sexual Function Index (OmtFSFI) score, from 18 (best) to 72 (worst)
Post-operative issues | Instantly, 6 months and 24 months
  Epidemiologic census of post-operative issues

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No